CLINICAL TRIAL: NCT02226341
Title: Open-label Prospective Randomized Study to Determine the Efficacy and Safety of Two Dosing Regimens of ACTHar in the Treatment of Proliferative Lupus Nephritis.
Brief Title: ACTHar in the Treatment of Lupus Nephritis
Acronym: ACTHar
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Anca Askanase, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAN4752
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Lupus Nephritis
Keywords: Lupus; Lupus Nephritis; ACTHar; Columbia; Rheumatology; CUMC; Autoimmune; SLE; Proliferative Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CellCept daily & ACTHar gel biw (Active Comparator): Patients will be treated with CellCept 3 grams daily and ACTHar gel 80 U biw for 3 months per Aim 1. After 3 months, patients with complete response will stop ACTHar gel but continue CellCept 3 grams daily for another 3 months whereas patients with partial response will continue CellCept 3 grams daily and be offered the option to continue ACTHar 80 U biw for another 3 months. After 6 months, all patients will continue CellCept at a dose of 2 grams daily for another 18 months.
  Interventions: Drug: CellCept; Drug: ACTHar gel
- CellCept daily & ACTHar gel qod (Active Comparator): Patients will be treated with CellCept 3 grams daily for 3 months, and ACTHar gel 80 U qod for the first month and ACTHar gel 80 U biw for the following 2 months per Aim 2. After 3 months, patients with complete response will stop ACTHar gel but continue CellCept 3 grams daily for another 3 months whereas patients with partial response will continue CellCept 3 grams daily and be offered the option to continue ACTHar 80 U biw for another 3 months. After 6 months, all patients will continue CellCept at a dose of 2 grams daily for another 18 months.
  Interventions: Drug: CellCept; Drug: ACTHar gel

INTERVENTIONS:
Drug: CellCept — For both arms:
  CellCept 3 grams daily, oral, from Week 0-24 CellCept 2 grams daily, oral, from Week 25-144
  Other Names: Mycophenolate Mofetil
Drug: ACTHar gel — Arm 1: 80 U biw, subcutaneous, for 3 months. Optionally additional 3 months of 80 U biw if a patient has partial response.
  Arm 2: 80 U qod, subcutaneous, for 1 month, then 80 U biw, subcutaneous, for 2 months. Optionally additional 3 months of 80 U biw if a patient has partial response.
  Other Names: ACTHar; H.P. ACTHar Gel; Repository corticotropin

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a disease in which the immune system attacks the healthy cells and tissues, causing inflammation that can damage organs in the body. About 50% of SLE patients experience inflammation in the kidneys. The purpose of this study is to determine the effectiveness and safety of two dosing arms of ACTHar gel in treating proliferative Lupus Nephritis (LN). This study hypothesizes that both dosing arms of ACTHar are safe and effective in treating proliferative LN (Class III and IV).

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is an autoimmune disease of unknown etiology that mainly affects females of childbearing age. The disease is characterized by immune activation and the development of autoantibodies.

About 50% of SLE patients experience inflammation of the kidneys. Lupus Nephritis (LN) is a major cause of morbidity and mortality in patients with SLE. Mycophenolate Mofetil (MMF), accompanied by Prednisone, is considered the current standard of care for LN. However, long-term use of Prednisone has many serious side effects.

ACTHar Gel is an FDA approved drug comprised of an active substance called adrenocorticotropic hormone (ACTH). ACTH belongs to an anti-inflammatory group called melanocortins and carries out its effects by binding to five different melanocortin receptors (MCRs). Specifically, ACTH binding to melanocortin 2 receptor subtype (MC2R) on the adrenal cortex stimulates the production of cortisol that reduces inflammation in the kidney. In addition to binding to melanocortin 1-5 receptor subtype (MC1-5R) and acting directly on kidney tissues, ACTH may bind to MCRs on various cell types, such as immune cells, and activate processes to protect the kidney.

This study will evaluate the most effective dose of ACTHar gel in proliferative LN (Class III and IV) when given with MMF, the standard of care LN therapy. The intent of this study is to determine the effectiveness and safety of ACTHar gel in an attempt to change the clinical care requirements regarding steroid use in treating LN.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Systemic Lupus Erythematosus (SLE) by American College of Rheumatology (ACR)/SLICC criteria
2. Age ≥ 16 years
3. Active lupus nephritis defined by:

   a. Kidney biopsy documentation of International Society of Nephrology/Renal Pathology Society (ISN/RPS) Class III or Class IV proliferative nephritis (including Class V occurring in combination with Class III or IV) within 12 months and a urine protein/creatinine ratio >1 at time of entry to study
4. Ability to provide informed consent

Exclusion Criteria:

1. Moderately severe anemia (Hgb < 8 mg/dL)
2. Neutropenia (< 1,000/mm3)
3. Thrombocytopenia (platelets < 50,000/mm3)
4. Positive purified protein derivative (PPD) test confirmed by positive Quantiferon TB gold.
5. Pulmonary fibrotic changes on chest radiograph consistent with prior healed tuberculosis
6. Active infections that in the opinion of the investigator increase the risks to the subject.
7. Known human immunodeficiency virus (HIV) and hepatitis B or C
8. End-stage renal disease (estimated GFR clearance < 20 mL/min/1.73 m2)
9. History of cancer, except carcinoma in situ and treated basal and squamous cell carcinomas
10. Pregnancy
11. Lactation
12. Unwillingness to use a medically acceptable form of birth control (including but not limited to a diaphragm, an intrauterine device, progesterone implants or injections, oral contraceptives, the double-barrier method, or a condom)
13. Previous failure to respond to MMF
14. Use of rituximab within the past year
15. Use of experimental therapeutic agents within the past 60 days
16. Greater than or equal to 5 times the upper limit of normal of liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], or alkaline phosphatase)
17. Severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease (or, in the investigator's opinion, any other concomitant medical condition that places the participant at risk by participating in this study) with the exception of diseases or conditions related to active SLE
18. Current substance abuse

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anca D Askanase, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University - Herbert Irving Pavilion, New York, New York, United States

REFERENCES:
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Lam GK, Petri M. Assessment of systemic lupus erythematosus. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S120-32. PMID 16273796
- [Background] Austin HA 3rd, Muenz LR, Joyce KM, Antonovych TT, Balow JE. Diffuse proliferative lupus nephritis: identification of specific pathologic features affecting renal outcome. Kidney Int. 1984 Apr;25(4):689-95. doi: 10.1038/ki.1984.75. PMID 6482173
- [Background] Weening JJ, D'Agati VD, Schwartz MM, Seshan SV, Alpers CE, Appel GB, Balow JE, Bruijn JA, Cook T, Ferrario F, Fogo AB, Ginzler EM, Hebert L, Hill G, Hill P, Jennette JC, Kong NC, Lesavre P, Lockshin M, Looi LM, Makino H, Moura LA, Nagata M; International Society of Nephrology Working Group on the Classification of Lupus Nephritis; Renal Pathology Society Working Group on the Classification of Lupus Nephritis. The classification of glomerulonephritis in systemic lupus erythematosus revisited. Kidney Int. 2004 Feb;65(2):521-30. doi: 10.1111/j.1523-1755.2004.00443.x. PMID 14717922
- [Background] Bomback AS, Canetta PA, Beck LH Jr, Ayalon R, Radhakrishnan J, Appel GB. Treatment of resistant glomerular diseases with adrenocorticotropic hormone gel: a prospective trial. Am J Nephrol. 2012;36(1):58-67. doi: 10.1159/000339287. Epub 2012 Jun 19. PMID 22722778
- [Background] Schweitzer EJ, Yoon S, Fink J, Wiland A, Anderson L, Kuo PC, Lim JW, Johnson LB, Farney AC, Weir MR, Bartlett ST. Mycophenolate mofetil reduces the risk of acute rejection less in African-American than in Caucasian kidney recipients. Transplantation. 1998 Jan 27;65(2):242-8. doi: 10.1097/00007890-199801270-00017. PMID 9458022
- [Background] Dooley MA, Jayne D, Ginzler EM, Isenberg D, Olsen NJ, Wofsy D, Eitner F, Appel GB, Contreras G, Lisk L, Solomons N; ALMS Group. Mycophenolate versus azathioprine as maintenance therapy for lupus nephritis. N Engl J Med. 2011 Nov 17;365(20):1886-95. doi: 10.1056/NEJMoa1014460. PMID 22087680
- [Background] Belmont HM, Levartovsky D, Goel A, Amin A, Giorno R, Rediske J, Skovron ML, Abramson SB. Increased nitric oxide production accompanied by the up-regulation of inducible nitric oxide synthase in vascular endothelium from patients with systemic lupus erythematosus. Arthritis Rheum. 1997 Oct;40(10):1810-6. doi: 10.1002/art.1780401013. PMID 9336415
- See also: CUMC Rheumatology Research Website — http://www.rheumatologyatcolumbia.org/index-3.html

RESULTS

PARTICIPANT FLOW:
Groups:
- CellCept Daily & ACTHar Gel BIW (Two Times Per Week): Patients will be treated with CellCept 3 grams daily and ACTHar gel 80 U BIW for 3 months per Aim 1. After 3 months, patients with complete response will stop ACTHar gel but continue CellCept 3 grams daily for another 3 months whereas patients with partial response will continue CellCept 3 grams daily and be offered the option to continue ACTHar 80 U biw for another 3 months. After 6 months, all patients will continue CellCept at a dose of 2 grams daily for another 18 months.
- CellCept Daily & ACTHar Gel TIW (Three Times Per Week): Patients will be treated with CellCept 3 grams daily for 3 months, and ACTHar gel 80 U TIW for the first month and ACTHar gel 80 U BIW for the following 2 months per Aim 2. After 3 months, patients with complete response will stop ACTHar gel but continue CellCept 3 grams daily for another 3 months whereas patients with partial response will continue CellCept 3 grams daily and be offered the option to continue ACTHar 80 U BIW for another 3 months. After 6 months, all patients will continue CellCept at a dose of 2 grams daily for another 18 months.
Period: Overall Study
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.5 [22 to 36] | 28.5 [24 to 34] | 26.5 [23.5 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Complete Response (CR)
Description: Complete response (CR) is defined as all of the following criteria having been achieved:
  1. Stabilization of estimated glomerular filtration rate (eGFR) (i.e., a 6-month eGFR level ± 10% of baseline) or improvement if the screening value is changed from patient's baseline
  2. Inactive urinary sediment (red blood cells per high-power field [RBCs/HPF] < 5-10, not due to gyn bleeding)
  3. Urine protein/creatinine ratio < 0.5
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 4 | 4
Participants | 2 | 0

2. Secondary Outcome: Number of Responders
Description: Responders = Complete Responders (CR) + Partial Responders (PR). PR = improvement from baseline of at least ≥ 50% in all abnormal renal parameters (proteinuria and serum creatinine) without deterioration of any measurements at 6 months
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 4 | 4
Participants | 2 | 1

3. Secondary Outcome: Number of Patients With Extra-renal Flares
Description: Frequency of extra-renal flares as defined by the SELENA-SLEDAI Flare Index. Extra-renal disease activity measured by SELENA-SLEDAI and BILAG
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 4 | 4
Participants | 0 | 1

4. Secondary Outcome: Number of Patients With Steroid -Like Side Effects
Description: Steroid -like side effects: increase in blood pressure (BP) by 20 mmHg for both systolic blood pressure (SBP) and diastolic blood pressure (DBP), increased blood sugar with a fasting plasma glucose level ≥ 126 mg/dl, weight gain ≥ 10% of the initial weight, infections
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

5. Secondary Outcome: Number of Patients With Side Effects
Description: Number of participants who experienced side effects from taking ACTHar
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

6. Other Pre Specified Outcome: Mean Urinary Lymphocytes
Description: Urinary markers of active inflammatory nephritis
Time Frame: Upon study completion, up to 30 months
Population: Data was not collected due to lack of funding leading to early termination of the study.
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Mean Cortisol Levels
Description: Cortisol levels 8 hours after ACTHar dose in 2-3 patients per dosing arm
Time Frame: Upon study completion, up to 30 months
Population: Data was not collected due to lack of funding leading to early termination of the study.
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) (N=4) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week) (N=4)
Extra-renal flare (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CellCept Daily & ACTHar Gel BIW (Two Times Per Week) (N=4) | CellCept Daily & ACTHar Gel TIW (Three Times Per Week) (N=4)
Renal flare (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02226341/Prot_SAP_000.pdf